CLINICAL TRIAL: NCT06566482
Title: Mini-dose Dexmedetomidine-Esketamine Supplemented Analgesia for Postoperative Sleep Promotion in Patients at High-risk of Obstructive Sleep Apnea: A Randomized Trial
Brief Title: Mini-dose Dexmedetomidine-Esketamine Supplemented Analgesia in Patients at High-risk of OSA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anesthesiology, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2024-234
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Obstructive Sleep Apnea; Surgery; Dexmedetomidine; Esketamine; Postoperative Sleep Quality
Keywords: Obstructive Sleep Apnea; Surgery; Dexmedetomidine; Esketamine; Postoperative sleep quality
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine-esketamine combination (Experimental): Patient-controlled analgesia is established with dexmedetomidine (1 μg/ml), esketamine (1 mg/ml), and sufentanil (1 μg/ml) in a total volume of 100 ml. The pump is programmed to deliver 2-ml boluses at 6 to 8-minute lockout intervals with a background infusion rate at 1 ml/h. Patient-controlled analgesia is provided for at least 24 hours but no more than 48 hours after surgery.
  Interventions: Drug: Dexmedetomidine-esketamine combination
- Placebo (Placebo Comparator): Patient-controlled analgesia is established with sufentanil (1 μg/ml) in a total volume of 100 ml. The pump is programmed to deliver 2-ml boluses at 6 to 8-minute lockout intervals with a background infusion rate at 1 ml/h. Patient-controlled analgesia is provided for at least 24 hours but no more than 48 hours after surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine-esketamine combination — Patient-controlled analgesia is established with dexmedetomidine (1 μg/ml), esketamine (1 mg/ml), and sufentanil (1 μg/ml) in a total volume of 100 ml. The pump is programmed to deliver 2-ml boluses at 6 to 8-minute lockout intervals with a background infusion rate at 1 ml/h. Patient-controlled analgesia is provided for at least 24 hours but no more than 48 hours after surgery.
  Other Names: Dexmedetomidine-esketamine group
  Arms: Dexmedetomidine-esketamine combination
Drug: Placebo — Patient-controlled analgesia is established with sufentanil (1 μg/ml) in a total volume of 100 ml. The pump is programmed to deliver 2-ml boluses at 6 to 8-minute lockout intervals with a background infusion rate at 1 ml/h. Patient-controlled analgesia is provided for at least 24 hours but no more than 48 hours after surgery.
  Other Names: Placebo group
  Arms: Placebo

SUMMARY:
Patients with obstructive sleep apnea (OSA) are at increased risk of developing sleep disturbances after surgery. Dexmedetomidine is a highly selective α2-adrenergic agonist with sedative, analgesic, and anxiolytic effects. Ketamine is a noncompetitive N-methyl-d-aspartate (NMDA) receptor antagonist. Esketamine is the S-enantiomer of racemic ketamine and twice as potent as racemic ketamine for analgesia. A recent trial showed that mini-dose esketamine-dexmedetomidine in combination with opioids improved analgesia and subjective sleep quality after scoliosis correction surgery. This trial is designed to test the hypothesis that mini-dose dexmedetomidine-esketamine supplemented analgesia may improve postoperative sleep quality in patients at high-risk of OSA.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is characterized by repetitive narrowing or obstruction of the upper airway during sleep, resulting in recurrent hypoxemia and hypercapnia and disordered sleep. During the postoperative period, the residual effects of anesthetics, sedatives, analgesics, and muscle relaxants suppress the activation of airway muscles; surgical stress, pain, and environmental interference further deteriorate sleep quality. All these factors aggravate the pathophysiological changes in OSA patients and may lead to worse perioperative outcomes, including increased respiratory and cardiac events, intensive care unit (ICU) admission and delirium, as well as prolonged length of hospital stay.

Opioids are commonly used for postoperative analgesia. Patients with OSA have significantly increased sensitivity to the side effects of opioids, such as central respiratory depression (reduced central respiratory drive) and peripheral respiratory depression (airway collapse). Opioids themselves can also cause sleep disturbances, as manifested by sleep fragmentation, decreased rapid-eye-movement sleep, and frequent nightmares. On the other hand, sleep deprivations can also lead to increased pain sensitivity and thus opioid consumption. Therefore, it is important to explore better postoperative analgesia to improve postoperative sleep quality of patients at high-risk of OSA.

Dexmedetomidine is a highly selective α2-adrenergic agonist with sedative, analgesic, and anxiolytic effects. It produces sedation by activating the endogenous sleep-promoting pathway and produces a state resembling nonrapid eye movement sleep. Ketamine is a noncompetitive N-methyl-d-aspartate (NMDA) receptor antagonist. When given in sub-anaesthetic doses, ketamine produces analgesic and anti-hyperalgesic effects and is recommended as a component of multimodal analgesia. Esketamine is the S-enantiomer of racemic ketamine and approximately twice as potent as racemic ketamine for analgesia.

A recent trial showed that mini-dose esketamine-dexmedetomidine in combination with opioids improved analgesia and subjective sleep quality after scoliosis correction surgery. This trial is designed to test the hypothesis that mini-dose dexmedetomidine-esketamine supplemented analgesia may improve sleep quality in patients at high-risk of OSA after thoracic or abdominal surgery.

ELIGIBILITY:
Inclusion criteria:

1. Aged ≥18 years but ≤80 years;
2. Preoperative diagnosis of OSA, or judged to be at moderate-to-high risk of OSA according to the STOP-Bang Questionnaire;
3. Scheduled to undergo thoracoscopic or laparoscopic surgery under general anesthesia, with an expected surgical duration of ≥1 hours, and required patient-controlled intravenous analgesia (PCIA) after surgery.

Exclusion criteria:

1. Diagnosed as central sleep apnea syndrome;
2. Previous history of schizophrenia, epilepsy, Parkinson disease, or myasthenia gravis.
3. History of schizophrenia, or having antipsychotic drugs (including antidepressants or anxiolytics);
4. Inability to communicate in the preoperative period because of coma, profound dementia, or deafness;
5. History of drug or alcohol dependence, or sedative or hypnotic therapy within 1 month before surgery;
6. Contraindications to ketamine (such as hyperthyroidism, pheochromocytoma, or glaucoma);
7. Sick sinus syndrome, severe sinus bradycardia (<50 beats per minute), or second-degree or above atrioventricular block without pacemaker;
8. Contraindications to high-flow nasal cannula therapy (such as mediastinal emphysema, shock or hypotension, cerebrospinal fluid leakage, nasosinusitis, otitis media, or deviation of nasal septum);
9. Severe hepatic dysfunction (Child-Pugh class C), severe renal dysfunction (requirement of renal replacement therapy), severe heart dysfunction (preoperative New York Heart Association functional classification ≥3 or left ventricular ejection fraction <30%), or ASA classification IV or above;
10. Expected intensive care unit (ICU) admission with tracheal intubation after surgery;
11. Other conditions that are considered unsuitable for study participation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Subjective sleep quality during the first night after surgery. | During the first night after surgery.
  Subjective sleep quality is assessed with the Richards-Campbell Sleep Questionnaire (RCSQ). The RCSQ is a self-reported measure of subjective sleep quality with 5 items, including sleep depth, sleep latency, awakening, return to sleep, and overall sleep quality; the score of each item ranges from 0 to 100, with a higher score indicating better sleep.

SECONDARY OUTCOMES:
Sleep structure parameters during the first night after surgery. | During the first night after surgery
  Sleep structure is monitored with a polysomnograph from 9:00 pm on the night of surgery to 6:00 am the next morning. Sleep stages and respiratory events are scored according to the American Academy of Sleep Medicine (AASM) manual by qualified sleep physicians.
Cumulative subjective sleep quality score after surgery | During the first three nights after surgery.
  Subjective sleep quality is assessed with the Richards-Campbell Sleep Questionnaire (RCSQ). The RCSQ is a self-reported measure of subjective sleep quality with 5 items, including sleep depth, sleep latency, awakening, return to sleep, and overall sleep quality; the score of each item ranges from 0 to 100, with a higher score indicating better sleep.
Proportion of patients with poor sleep quality after surgery. | During the first three nights after surgery.
  Subjective sleep quality is assessed with the Richards-Campbell Sleep Questionnaire (RCSQ). Poor sleep quality is defined as overall RCSQ<50 on any night after surgery.
Area under curve of pain intensity score within 3 days after surgery. | Up to 3 days after surgery.
  Pain intensity is assessed twice daily (8-10 am and 18-20 pm) with the numeric rating scale (NRS), an 11-point scale where 0=no pain and 10=the worst pain.
Subjective sleep quality at 30 days after surgery. | At 30 days after surgery.
  Subjective sleep quality is assessed with the Pittsburgh Sleep Quality Index (PSQI; score ranges from 0 to 21, with higher score indicating worse sleep quality).

OTHER OUTCOMES:
Sedation level within 3 days after surgery. | Up to 3 days after surgery.
  Sedation level is assessed at 2 hours and twice daily (8-10 am and 18-20 pm) after surgery with the Richmond Agitation Sedation Scale (RASS), with scores ranging from -5(unarousable) to +4 (combative) and 0 indicates alert and calm.
Length of stay in hospital after surgery. | Up to 30 days after surgery.
  Length of stay in hospital after surgery.
Incidence of delayed neurocognitive recovery. | At 30 days after surgery.
  Cognitive function is assessed with the Telephone Montreal Cognitive Assessment (T-MoCA; scores range from 0 to 22, with higher score indicating better function) before surgery and at 30 days after surgery. A T-MoCA score reduction of 1 standard deviation (SD) or more from baseline is defined the occurrence of delayed neurocognitive recovery.
Incidence of major complications after surgery. | Up to 30 days after surgery.
  Major complications are defined as new-onset medical events that are deemed harmful and require therapeutic intervention, that is grade II or higher on the Clavien-Dindo classification.
All-cause 30-day mortality. | Up to 30 days after surgery.
  All-cause 30-day mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, M.D., Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gottlieb DJ, Punjabi NM. Diagnosis and Management of Obstructive Sleep Apnea: A Review. JAMA. 2020 Apr 14;323(14):1389-1400. doi: 10.1001/jama.2020.3514. PMID 32286648
- [Background] Benjafield AV, Ayas NT, Eastwood PR, Heinzer R, Ip MSM, Morrell MJ, Nunez CM, Patel SR, Penzel T, Pepin JL, Peppard PE, Sinha S, Tufik S, Valentine K, Malhotra A. Estimation of the global prevalence and burden of obstructive sleep apnoea: a literature-based analysis. Lancet Respir Med. 2019 Aug;7(8):687-698. doi: 10.1016/S2213-2600(19)30198-5. Epub 2019 Jul 9. PMID 31300334
- [Background] Young T, Evans L, Finn L, Palta M. Estimation of the clinically diagnosed proportion of sleep apnea syndrome in middle-aged men and women. Sleep. 1997 Sep;20(9):705-6. doi: 10.1093/sleep/20.9.705. PMID 9406321
- [Background] Kapur VK, Auckley DH, Chowdhuri S, Kuhlmann DC, Mehra R, Ramar K, Harrod CG. Clinical Practice Guideline for Diagnostic Testing for Adult Obstructive Sleep Apnea: An American Academy of Sleep Medicine Clinical Practice Guideline. J Clin Sleep Med. 2017 Mar 15;13(3):479-504. doi: 10.5664/jcsm.6506. PMID 28162150
- [Background] Brown KA. Intermittent hypoxia and the practice of anesthesia. Anesthesiology. 2009 Apr;110(4):922-7. doi: 10.1097/ALN.0b013e31819c480a. PMID 19293703
- [Background] Chung F, Liao P, Yegneswaran B, Shapiro CM, Kang W. Postoperative changes in sleep-disordered breathing and sleep architecture in patients with obstructive sleep apnea. Anesthesiology. 2014 Feb;120(2):287-98. doi: 10.1097/ALN.0000000000000040. PMID 24158049
- [Background] Hai F, Porhomayon J, Vermont L, Frydrych L, Jaoude P, El-Solh AA. Postoperative complications in patients with obstructive sleep apnea: a meta-analysis. J Clin Anesth. 2014 Dec;26(8):591-600. doi: 10.1016/j.jclinane.2014.05.010. Epub 2014 Oct 16. PMID 25439403
- [Background] Sun X, Yu J, Luo J, Xu S, Yang N, Wang Y. Meta-analysis of the association between obstructive sleep apnea and postoperative complications. Sleep Med. 2022 Mar;91:1-11. doi: 10.1016/j.sleep.2021.11.019. Epub 2022 Feb 11. PMID 35231774
- [Background] Lam KK, Kunder S, Wong J, Doufas AG, Chung F. Obstructive sleep apnea, pain, and opioids: is the riddle solved? Curr Opin Anaesthesiol. 2016 Feb;29(1):134-40. doi: 10.1097/ACO.0000000000000265. PMID 26545144
- [Background] Robertson JA, Purple RJ, Cole P, Zaiwalla Z, Wulff K, Pattinson KT. Sleep disturbance in patients taking opioid medication for chronic back pain. Anaesthesia. 2016 Nov;71(11):1296-1307. doi: 10.1111/anae.13601. Epub 2016 Aug 22. PMID 27545291
- [Background] Finan PH, Goodin BR, Smith MT. The association of sleep and pain: an update and a path forward. J Pain. 2013 Dec;14(12):1539-52. doi: 10.1016/j.jpain.2013.08.007. PMID 24290442
- [Background] Mo Y, Zimmermann AE. Role of dexmedetomidine for the prevention and treatment of delirium in intensive care unit patients. Ann Pharmacother. 2013 Jun;47(6):869-76. doi: 10.1345/aph.1AR708. PMID 23719785
- [Background] Nelson LE, Lu J, Guo T, Saper CB, Franks NP, Maze M. The alpha2-adrenoceptor agonist dexmedetomidine converges on an endogenous sleep-promoting pathway to exert its sedative effects. Anesthesiology. 2003 Feb;98(2):428-36. doi: 10.1097/00000542-200302000-00024. PMID 12552203
- [Background] Wu Y, Ma R, Zhou Q, Lau HY, Wang Y, Li J, Wen W. Dexmedetomidine-induced polysomnography as a diagnostic method in obstructive sleep apnea: a reliable alternative method? Sleep Med. 2021 Mar;79:145-151. doi: 10.1016/j.sleep.2021.01.005. Epub 2021 Jan 5. PMID 33524840
- [Background] Guldenmund P, Vanhaudenhuyse A, Sanders RD, Sleigh J, Bruno MA, Demertzi A, Bahri MA, Jaquet O, Sanfilippo J, Baquero K, Boly M, Brichant JF, Laureys S, Bonhomme V. Brain functional connectivity differentiates dexmedetomidine from propofol and natural sleep. Br J Anaesth. 2017 Oct 1;119(4):674-684. doi: 10.1093/bja/aex257. PMID 29121293
- [Background] Wu XH, Cui F, Zhang C, Meng ZT, Wang DX, Ma J, Wang GF, Zhu SN, Ma D. Low-dose Dexmedetomidine Improves Sleep Quality Pattern in Elderly Patients after Noncardiac Surgery in the Intensive Care Unit: A Pilot Randomized Controlled Trial. Anesthesiology. 2016 Nov;125(5):979-991. doi: 10.1097/ALN.0000000000001325. PMID 27571256
- [Background] Su X, Meng ZT, Wu XH, Cui F, Li HL, Wang DX, Zhu X, Zhu SN, Maze M, Ma D. Dexmedetomidine for prevention of delirium in elderly patients after non-cardiac surgery: a randomised, double-blind, placebo-controlled trial. Lancet. 2016 Oct 15;388(10054):1893-1902. doi: 10.1016/S0140-6736(16)30580-3. Epub 2016 Aug 16. PMID 27542303
- [Background] Zhang ZF, Su X, Zhao Y, Zhong CL, Mo XQ, Zhang R, Wang K, Zhu SN, Shen YE, Zhang C, Wang DX. Effect of mini-dose dexmedetomidine supplemented intravenous analgesia on sleep structure in older patients after major noncardiac surgery: A randomized trial. Sleep Med. 2023 Feb;102:9-18. doi: 10.1016/j.sleep.2022.12.006. Epub 2022 Dec 20. PMID 36587547
- [Background] Li HJ, Li CJ, Wei XN, Hu J, Mu DL, Wang DX. Dexmedetomidine in combination with morphine improves postoperative analgesia and sleep quality in elderly patients after open abdominal surgery: A pilot randomized control trial. PLoS One. 2018 Aug 14;13(8):e0202008. doi: 10.1371/journal.pone.0202008. eCollection 2018. PMID 30106963
- [Background] Parvizrad R, Nikfar S. Low-dose ketamine as an analgesic agent in the emergency department: Efficacy and safety. J Family Med Prim Care. 2022 Oct;11(10):6464-6471. doi: 10.4103/jfmpc.jfmpc_511_22. Epub 2022 Oct 31. PMID 36618192
- [Background] Brinck EC, Tiippana E, Heesen M, Bell RF, Straube S, Moore RA, Kontinen V. Perioperative intravenous ketamine for acute postoperative pain in adults. Cochrane Database Syst Rev. 2018 Dec 20;12(12):CD012033. doi: 10.1002/14651858.CD012033.pub4. PMID 30570761
- [Background] Schwenk ES, Viscusi ER, Buvanendran A, Hurley RW, Wasan AD, Narouze S, Bhatia A, Davis FN, Hooten WM, Cohen SP. Consensus Guidelines on the Use of Intravenous Ketamine Infusions for Acute Pain Management From the American Society of Regional Anesthesia and Pain Medicine, the American Academy of Pain Medicine, and the American Society of Anesthesiologists. Reg Anesth Pain Med. 2018 Jul;43(5):456-466. doi: 10.1097/AAP.0000000000000806. PMID 29870457
- [Background] Molero P, Ramos-Quiroga JA, Martin-Santos R, Calvo-Sanchez E, Gutierrez-Rojas L, Meana JJ. Antidepressant Efficacy and Tolerability of Ketamine and Esketamine: A Critical Review. CNS Drugs. 2018 May;32(5):411-420. doi: 10.1007/s40263-018-0519-3. PMID 29736744
- [Background] Moore TJ, Alami A, Alexander GC, Mattison DR. Safety and effectiveness of NMDA receptor antagonists for depression: A multidisciplinary review. Pharmacotherapy. 2022 Jul;42(7):567-579. doi: 10.1002/phar.2707. Epub 2022 Jun 26. PMID 35665948
- [Background] Qiu D, Wang XM, Yang JJ, Chen S, Yue CB, Hashimoto K, Yang JJ. Effect of Intraoperative Esketamine Infusion on Postoperative Sleep Disturbance After Gynecological Laparoscopy: A Randomized Clinical Trial. JAMA Netw Open. 2022 Dec 1;5(12):e2244514. doi: 10.1001/jamanetworkopen.2022.44514. PMID 36454569
- [Background] Duncan WC, Sarasso S, Ferrarelli F, Selter J, Riedner BA, Hejazi NS, Yuan P, Brutsche N, Manji HK, Tononi G, Zarate CA. Concomitant BDNF and sleep slow wave changes indicate ketamine-induced plasticity in major depressive disorder. Int J Neuropsychopharmacol. 2013 Mar;16(2):301-11. doi: 10.1017/S1461145712000545. Epub 2012 Jun 7. PMID 22676966
- [Background] Guo J, Qiu D, Gu HW, Wang XM, Hashimoto K, Zhang GF, Yang JJ. Efficacy and safety of perioperative application of ketamine on postoperative depression: A meta-analysis of randomized controlled studies. Mol Psychiatry. 2023 Jun;28(6):2266-2276. doi: 10.1038/s41380-023-01945-z. Epub 2023 Jan 20. PMID 36670198
- [Background] Gregoire C, De Kock M, Henrie J, Cren R, Lavand'homme P, Penaloza A, Verschuren F. Procedural Sedation With Dexmedetomidine in Combination With Ketamine in the Emergency Department. J Emerg Med. 2022 Aug;63(2):283-289. doi: 10.1016/j.jemermed.2022.01.017. Epub 2022 May 9. PMID 35550843
- [Background] Zhang Y, Cui F, Ma JH, Wang DX. Mini-dose esketamine-dexmedetomidine combination to supplement analgesia for patients after scoliosis correction surgery: a double-blind randomised trial. Br J Anaesth. 2023 Aug;131(2):385-396. doi: 10.1016/j.bja.2023.05.001. Epub 2023 Jun 9. PMID 37302963
- [Background] Chen L, He W, Liu X, Lv F, Li Y. Application of opioid-free general anesthesia for gynecological laparoscopic surgery under ERAS protocol: a non-inferiority randomized controlled trial. BMC Anesthesiol. 2023 Jan 27;23(1):34. doi: 10.1186/s12871-023-01994-5. PMID 36707777
- [Background] Nagappa M, Wong J, Singh M, Wong DT, Chung F. An update on the various practical applications of the STOP-Bang questionnaire in anesthesia, surgery, and perioperative medicine. Curr Opin Anaesthesiol. 2017 Feb;30(1):118-125. doi: 10.1097/ACO.0000000000000426. PMID 27898430